CLINICAL TRIAL: NCT06375291
Title: Which is More Effective for Pregnancy-Related Carpal Tunnel Syndrome? Ultrasound Guided Steroid İnjection, Splint, or Both
Brief Title: Pregnancy-Related Carpal Tunnel Syndrome Treatment
Status: Completed | Type: Observational
Sponsor: Mersin Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Suna Aşkın Turan, principle investigator, Pain Department Physician, Mersin Training and Research Hospital
Other Study IDs: MersinTRHpregcts
Record Dates: First submitted 2024-04-11; First posted 2024-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome Pregnancy
Keywords: carpal tunnel syndrome; pregnancy; steroid injection; ultrasound guided; splinting; Boston Carpal Tunnel Questionneaire; postpartum depression
MeSH Terms: conditions — Carpal Tunnel Syndrome; Depression, Postpartum | interventions — Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Steroid injected: The pregnant women with steroid injection
  Interventions: Other: splint /steroid injection/both
- 2: splint: The pregnant women with splinting
  Interventions: Other: splint /steroid injection/both
- 3:both: The pregnant women with steroid injection and splinting
  Interventions: Other: splint /steroid injection/both

INTERVENTIONS:
Other: splint /steroid injection/both — pregnant women treated in pain department by splint /steroid injection/both

SUMMARY:
The current retrospective study aimed to compare the effectiveness of local steroid injection plus splinting with that of local steroid injection or splinting alone. To assess the primary outcome, The Boston Carpal Tunnel Symptom Severity Scale was used. The secondary aim was the efficacy of the treatment on the patient's function severity and depression assessed by The Boston Carpal Tunnel Symptom Function Scale Edinburgh Depression Scale.

DETAILED DESCRIPTION:
Pregnancy-related carpal tunnel syndrome (PRCTS) is the most frequent mononeuropathy during pregnancy. During pregnancy there is fluid retention, which leads to edema on the ligaments that form the roof of the tunnel this leads to nerve compression. PRCTS is usually bilateral and mostly develops in the third trimester of pregnancy when body fluid retention and weight gain reach the maximum. The developed PRCTS in the first or second trimester usually aggravates in the third trimester.

Pregnancy-related CTS usually has a benign prognosis. In a systematic review study conducted by Padua et al., >50% of the patients reported that the symptoms persisted even after one year of treatment, and approximately 30% of the patients still had the symptoms after three years.

Activity modification, edema control, and wrist splinting keep the wrist in a neutral position and provide symptomatic relief of PRCTS. Steroid injection may provide temporary symptom relief in many patients. Surgery is seldom indicated; however, it may be considered when the symptoms and functional impairments are severe, nonsurgical treatments are ineffective, and significant nerve compression is detected in the electrophysiological study.

The most frequent indication related to corticosteroid therapy is acute CTS, developed in the third trimester. Many studies showed the effectiveness of steroid injection on PRCTS assessed by the Boston Carpal Tunnel Questionnaire and electrophysiological results. However, when assessing physical health problems in general, and in pregnant women in particular, it is important to be aware of mental health problems. Patients who report chronic pain also experience problems in a range of psychological domains, such as depression, anxiety, and general emotional functioning. It was found that higher postpartum depression scores were related to persistent CTS symptoms at 12 months postpartum.

Splinting is an effective method for both pregnant and nonpregnant CTS usually given as a first-line therapy. In nonpregnant populations with CTS, ultrasound-guided steroid injection with splinting was found more effective than injection or splinting alone. But there is no literature on pregnant women searching the efficacy of splinting, steroid injection or both. The current study aimed to compare the effectiveness of local steroid injection plus splinting with that of local steroid injection or splinting alone for symptom severity. The secondary aim was the efficacy of the treatment on the patient's function severity and depression. Boston Carpal Tunnel Symptom Severity Scale assessed the primary outcome. Boston Carpal Tunnel Functional Severity Scale and Edinburgh Depression Scale assessed the secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women in the third trimester treated for mild to moderate PRCTS in the Pain Department between 1 January 2021 and 1 March 2023 and followed up in the first month of the postpartum period were included in the study.

All the patients were diagnosed by clinical findings and electrophysiological studies.

-

Exclusion Criteria:

Patients with a lack of data, or secondary causes like as diabetes mellitus, gestational diabetes mellitus, eclampsia, preeclampsia, thyroid disorders, arthropathies, trauma to the hand or wrist, cervical disc pathology, and prior history of CTS (such as recurrence or a CTS diagnosis before pregnancy) were excluded.

-

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: All pregnant women in the third trimester treated for mild to moderate PRCTS in the Pain Department between 1 January 2021 and 1 March 2023 and followed up in the first month of the postpartum period were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Symptom severity | Before the intervention and 1. month, 3. months after the intervention
  Boston Carpal Tunnel Syndrome Questionnaire Symptom Severity

SECONDARY OUTCOMES:
function severity | Before the intervention and 1. month, 3. months after the intervention
  Boston Carpal Tunnel Syndrome Questionnaire Symptom Severity
pregnancy and postpartum depression | Before the intervention and 1. month, 3. months after the intervention
  assesed by Edinburg Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Suna Aşkın Turan, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The Data and materials are available from the corresponding author upon reasonable request and are subject to ethical review.